CLINICAL TRIAL: NCT04522778
Title: Innovative Central Line Securement Device: Line Complications and Quality of Life in the Pediatric Population as Compared to Traditional Securement Device
Brief Title: Innovative Central Line Securement Device in the Pediatric Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet enrollment targets
Sponsor: Ryan St. Pierre-Hetz (Other)
Responsible Party: Sponsor-Investigator, Ryan St. Pierre-Hetz, Pediatric Emergency Medicine Attending, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY19010059
Record Dates: First submitted 2020-08-17; First posted 2020-08-21 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Central Line Complication; Central Line Infection; Central Line-Associated Infection; Central Line Sepsis; Short Gut Syndrome; Quality of Life; Pediatric Disorder
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Patients with central lines ages 0-18 years old who have never worn a wearable central line securement device (vest) will be eligible for the study. Half of the participants will be randomized to the device arm while the other half of participants will be randomized to the non-device arm. They will be block randomized based on age upon enrollment. Those in the device arm will be given two wearable central line securement devices and the investigators will encourage continuous wear. The study will follow participants prospectively for approximately one year (2020 - 2021).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Device (Experimental): Those in the device arm will be given two wearable central line securement devices and the investigators will encourage continuous wear throughout the duration of the study.
  Interventions: Device: Wearable Central Line Securement Device (Vest); Other: Traditional Securement Dressing
- Traditional Securement Dressing (Active Comparator): Those is the non-device arm will continue to wear a traditional central line securement dressing as is the standard of care.
  Interventions: Other: Traditional Securement Dressing

INTERVENTIONS:
Device: Wearable Central Line Securement Device (Vest) — The wearable central line securement device is a vest that has attachments for the central line to safely be secured to the body whether it is being used for infusion or unhooked. It also has a front flap, which protects the line from snagging on external objects.
  Arms: Device
Other: Traditional Securement Dressing — All subjects will use sterile dressings throughout the trial as this is the standard of care for central line securement. Subjects randomized to the dressing arm will continue to use standard of care sterile dressing as the only form of central line securement.

SUMMARY:
This study involves evaluating pediatric patients with central lines to determine differences in line complications and quality of life in those with a novel central line securement device (wrap) as compared to those who use a traditional securement device (dressing).

DETAILED DESCRIPTION:
Children with central lines experience line breaks, line dislodgment's and line infections as a result of traditional securement techniques (dressings). These issues lead to the patients' increased health care utilization and possibly to restriction of movement and delayed development as the children are restricted in their home environment. The purpose of this study is to determine if a wearable central line securement device, can decrease the number of line breaks, line dislodgment and line infections as compared to traditional securement techniques. Events per month would be calculated for each arm before and after intervention and analyzed for treatment effect. The hypothesis is that the use of this wearable central line securement device can reduce line breaks, line dislodgment and line infections as compared to the traditional adhesive dressing. A secondary outcome for evaluation will be quality of life. This will be analyzed with a standardized quality of life survey and treatment effect will be reported as an ordinal odds ratio. Children are naturally active, however their activity is restricted by the parents given the delicate nature of their line. This study looks to see if quality of life can be improved a more secure wearable attachment device, as compared to traditional securement techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a central line ages 0-18 years old who have never worn a wearable central line securement device (vest) will be eligible for the study.

Exclusion Criteria:

* Those children who currently wear a central line securement device (vest)
* Children with central lines who are 19 years or older
* Those females with central lines and Tanner 2 breast or greater breast development as a wearable central line securement device (vest) will not fit properly to secure the central line and may increase the risk of the central line complications.
* If the patient does develop breast during the time of the study then the patient will no longer wear the wrap and will go back to securing their device in the traditional way. The investgators will still collect data on that patient and they will be evaluated in the device arm consistent with the intention to treat principle.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Mazzarini, MD, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwang FR, Stavropoulos SW, Shlansky-Goldberg RD, Mondschein JI, Patel AA, Solomon JA, Itkin M, Soulen MC, Chittams JL, Trerotola SO. Tunneled infusion catheter breakage: frequency and repair kit outcomes. J Vasc Interv Radiol. 2008 Feb;19(2 Pt 1):201-6. doi: 10.1016/j.jvir.2007.08.030. PMID 18341949
- [Background] Lundgren IS, Zhou C, Malone FR, McAfee NG, Gantt S, Zerr DM. Central venous catheter repair is associated with an increased risk of bacteremia and central line-associated bloodstream infection in pediatric patients. Pediatr Infect Dis J. 2012 Apr;31(4):337-40. doi: 10.1097/INF.0b013e31823eeec5. PMID 22146741
- [Background] Cesaro S, Corro R, Pelosin A, Gamba P, Zadra N, Fusaro F, Pillon M, Cusinato R, Zampieri C, Magagna L, Cavaliere M, Tridello G, Zanon G, Zanesco L. A prospective survey on incidence and outcome of Broviac/Hickman catheter-related complications in pediatric patients affected by hematological and oncological diseases. Ann Hematol. 2004 Mar;83(3):183-8. doi: 10.1007/s00277-003-0796-9. Epub 2003 Nov 13. PMID 15064868
- [Background] Ullman AJ, Marsh N, Mihala G, Cooke M, Rickard CM. Complications of Central Venous Access Devices: A Systematic Review. Pediatrics. 2015 Nov;136(5):e1331-44. doi: 10.1542/peds.2015-1507. Epub 2015 Oct 12. PMID 26459655
- [Background] Peng C, Monagle P, Newall F. Clinical outcomes of management of CVAD occlusions. Arch Dis Child. 2011 Sep;96(9):885-7. doi: 10.1136/adc.2010.194969. Epub 2011 Mar 11. PMID 21398316
- [Background] Rey C, Alvarez F, De La Rua V, Medina A, Concha A, Diaz JJ, Menendez S, Los Arcos M, Mayordomo-Colunga J. Mechanical complications during central venous cannulations in pediatric patients. Intensive Care Med. 2009 Aug;35(8):1438-43. doi: 10.1007/s00134-009-1534-0. Epub 2009 Jun 16. PMID 19529913
- [Background] Winkler MF, DiMaria-Ghalili RA, Guenter P, Resnick HE, Robinson L, Lyman B, Ireton-Jones C, Banchik LH, Steiger E. Characteristics of a Cohort of Home Parenteral Nutrition Patients at the Time of Enrollment in the Sustain Registry. JPEN J Parenter Enteral Nutr. 2016 Nov;40(8):1140-1149. doi: 10.1177/0148607115586575. Epub 2015 May 13. PMID 25972431
- [Background] Burckhardt CS, Anderson KL. The Quality of Life Scale (QOLS): reliability, validity, and utilization. Health Qual Life Outcomes. 2003 Oct 23;1:60. doi: 10.1186/1477-7525-1-60. PMID 14613562
- [Background] Gimeno-Santos E, Raste Y, Demeyer H, Louvaris Z, de Jong C, Rabinovich RA, Hopkinson NS, Polkey MI, Vogiatzis I, Tabberer M, Dobbels F, Ivanoff N, de Boer WI, van der Molen T, Kulich K, Serra I, Basagana X, Troosters T, Puhan MA, Karlsson N, Garcia-Aymerich J; PROactive consortium. The PROactive instruments to measure physical activity in patients with chronic obstructive pulmonary disease. Eur Respir J. 2015 Oct;46(4):988-1000. doi: 10.1183/09031936.00183014. Epub 2015 May 28. PMID 26022965

RESULTS

PARTICIPANT FLOW:
Groups:
- Device: Those in the device arm will be given two wearable central line securement devices and the investigators will encourage continuous wear throughout the duration of the study. They will continued to wear sterile dressing, the standard of care, underneath the device.
  Wearable Central Line Securement Device (Vest): The wearable central line securement device is a vest that has attachments for the central line to safely be secured to the body whether it is being used for infusion or unhooked. It also has a front flap, which protects the line from snagging on external objects.
- Traditional Securement Dressing: Those is the non-device arm will continue to wear a traditional central line securement dressing as is the standard of care.
  Traditional Securement Dressing: This is a adhesive patch that is traditionally used to secure the external portion of a central line.
Period: Overall Study
Arm/Group | Device | Traditional Securement Dressing
Started | 12 | 11
Completed | 11 | 10
Not Completed | 1 | 1
Not completed — Patient did not want to wear the device | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Device: After randomization and device securementall families filled out a baseline demographics form and a baseline QOL survey. Patients were then followed for 12 months from initial enrollment. At subsequent clinic visits patients and families filled out follow-up surveys detailing potential line related complications. They were also given the same QOL survey that they filled out at the time of initial enrollment. These follow-up surveys were administered between 3-6 times throughout the year. Subjects' charts were routinely reviewed over the study, monitoring for ER visits, hospital admissions and line related complications.
- Traditional Securement Dressing: After randomization all families filled out a baseline demographics form and a baseline QOL survey. Patients were then followed for 12 months from initial enrollment. At subsequent clinic visits patients and families filled out follow-up surveys detailing potential line related complications. They were also given the same QOL survey that they filled out at the time of initial enrollment. These follow-up surveys were administered between 3-6 times throughout the year. Subjects' charts were routinely reviewed over the study, monitoring for ER visits, hospital admissions and line related complications.
- Total: Total of all reporting groups
Arm/Group | Device | Traditional Securement Dressing | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.99 (4.13) | 5.46 (5.16) | 5.21 (4.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 6 | 7 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome - Line Breaks
Description: Number of line breaks defined as any mechanical trauma to the line that required repair but not replacement of the line.
Time Frame: For a maximum of 1 year from enrollment
Measure: Mean (Standard Deviation); unit: Line breaks/month
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Line breaks/month | .05 (.09) | .05 (.07)
Statistical Analysis 1: Comparison: Device; A ratio of events per month was calculated for each participant. Participants were compared to themselves prior to intervention (i.e. event ratios pre intervention were compared to event ratios following intervention.); Test type: Other; p = .029, t-test, 1 sided

2. Primary Outcome: Primary Outcome - Line Replacement
Description: Number of line replacements in which a line was removed from the patient and a new line was placed.
Time Frame: For a maximum of 1 year from enrollment
Measure: Mean (Standard Deviation); unit: Events per month
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Events per month | .076 (.15) | .05 (.16)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .35, t-test, 1 sided

3. Primary Outcome: Primary Outcome - Line Infections
Description: Number of line infections defined as a positive blood culture drawn from a central line.
Time Frame: For a maximum of 1 year from enrollment
Measure: Mean (Standard Deviation); unit: Infections/Month
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Infections/Month | .086 (.12) | .075 (.12)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .334, t-test, 1 sided

4. Secondary Outcome: How Has the Vest or Dressing Affected Your Ability as a Family to Participate in Daily Activities?
Description: Survey modified from Baxter Scale of Quality of Life. These surveys were completed by family members or patients. Responses were recorded as a likert scale from 1-5 with 1 being much worse, 5 being much better. Quality of life data was recorded using ordinal scales. Therefore, we compared responses to individual questions between the dressing group and vest group using ordinal logistic regression, adjusting for clustering of responses within a participant. We present the mean and standard deviation for all responses as well as the ordinal odds ratio and 95% confidence intervals for a unit change in response level for each question.
Time Frame: Responses were recorded every Thursday follow up appointment, save for holidays between January 2021 and September 2022. The maximum number of responses of a participant was 5 over a maximum of 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 33 | 30
score on a scale | 3.82 (.982) | 2.875 (.712)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .005, Chi-squared; Odds Ratio (OR) = 38.26, 95% CI 2-sided [2.926154 to 500.4402], Standard Error of Mean 50.195

5. Secondary Outcome: How Has the Vest or Dressing Affected Your Child's Ability to be Active?
Description: as for outcome 4
Time Frame: Responses were recorded every Thursday follow up appointment, save for holidays between January 2021 and September 2022. The maximum number of responses for an individual was 5 over a 12 month period.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 22 | 36
score on a scale | 3.45 (1.06) | 3.78 (1.02)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .003, Chi-squared; Odds Ratio (OR) = 30.975, 95% CI 2-sided [3.22 to 297.17], Standard Error of Mean 35.73483

6. Secondary Outcome: How Has the Vest or Dressing Affected Your Child's Ability to Participate in Typical Activities With Peers or Siblings?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 36 | 31
score on a scale | 3.86 (1.10) | 2.74 (0.73)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .004, Chi-squared; Odds Ratio (OR) = 27.36, 95% CI 2-sided [2.82 to 265.45], Standard Error of Mean 31.72

7. Secondary Outcome: How Has the Vest or Dressing Affected Your Ability to Keep Your Child's Central Line Safe?
Description: Survey modified from Baxter Scale of Quality of Life. These surveys were completed by family members or patients. Responses were recorded as a likert scale from 1-5 with 1 being much worse, 5 being much better and 6 being non applicable. Quality of life data was recorded using ordinal scales. Therefore, we compared responses to individual questions between the dressing group and vest group using ordinal logistic regression, adjusting for clustering of responses within a participant. We present the mean and standard deviation for all responses as well as the ordinal odds ratio and 95% confidence intervals for a unit change in response level for each question.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 32 | 31
score on a scale | 4.03 (1.12) | 3.23 (0.80)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .011, Chi-squared; Odds Ratio (OR) = 10.93, 95% CI 2-sided [1.71 to 69.82], Standard Error of Mean 10.345

8. Secondary Outcome: Have You Been Worried About the Safety of Your Child's Central Line?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 43 | 32
score on a scale | 2.42 (1.2) | 2.84 (1.02)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .099, Chi-squared; Odds Ratio (OR) = .298, 95% CI 2-sided [.0706 to 1.258], Standard Error of Mean .2189

9. Secondary Outcome: Has Your Child Been Able to Take a Long Walk or Play?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 39 | 29
score on a scale | 3.37 (.82) | 3.41 (.87)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .312, Chi-squared; Odds Ratio (OR) = 1.201, 95% CI 2-sided [.549 to 6.562], Standard Error of Mean 1.201

10. Secondary Outcome: Has Your Child Been Able to Take a Short Walk Outside of the House?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 31 | 27
score on a scale | 3.68 (.79) | 3.52 (.89)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .753, Chi-squared; Odds Ratio (OR) = 1.519, 95% CI 2-sided [.112 to 20.623], Standard Error of Mean 2.022

11. Secondary Outcome: Are You Worried About Your Child's Current Health?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 31 | 19
score on a scale | 2.61 (0.99) | 2.74 (1.15)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .156, Chi-squared; Odds Ratio (OR) = .321, 95% CI 2-sided [.067 to 1.541], Standard Error of Mean .257

12. Secondary Outcome: Has Your Child Needed to Stay in Bed or a Chair During the Day?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 42 | 25
score on a scale | 1.19 (.51) | 1.4 (.76)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .318, Chi-squared; Odds Ratio (OR) = .458, 95% CI 2-sided [.099 to 2.122], Standard Error of Mean .358

13. Secondary Outcome: Has Your Child Needed Help With Eating, Dressing, Washing or Using the Toilet?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 42 | 25
score on a scale | 1.19 (.51) | 1.4 (.76)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .684, Chi-squared; Odds Ratio (OR) = .449, 95% CI 2-sided [.009 to 21.003], Standard Error of Mean .882

14. Secondary Outcome: Is Your Child Able to Socialize?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 40 | 26
score on a scale | 3.33 (.83) | 3.35 (1.02)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .460, Chi-squared; Odds Ratio (OR) = 2.335, 95% CI 2-sided [.246 to 22.194], Standard Error of Mean 2.683

15. Secondary Outcome: Is Your Child Able to do Sports/Exercise?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 34 | 20
score on a scale | 2.68 (1.01) | 2.85 (1.23)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .439, Chi-squared; Odds Ratio (OR) = 2.299, 95% CI 2-sided [.279 to 18.927], Standard Error of Mean 2.47293

16. Secondary Outcome: Is Your Child Able to Attend School/Pre-school?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 28 | 15
score on a scale | 2.96 (1.26) | 2.73 (1.33)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .714, Chi-squared; Odds Ratio (OR) = 1.634, 95% CI 2-sided [.119 to 22.514], Standard Error of Mean 2.187

17. Secondary Outcome: Does Having a Central Line Affect His/Her Participation in School?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 26 | 18
score on a scale | 2.11 (1.18) | 2.33 (1.28)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .412, Chi-squared; Odds Ratio (OR) = .379, 95% CI 2-sided [.037 to 3.842], Standard Error of Mean .448

18. Secondary Outcome: Does Having a Central Line Affect His or Her Learning at School?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 26 | 18
score on a scale | 1.5 (0.81) | 1.67 (1.03)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .558, Chi-squared; Odds Ratio (OR) = .579, 95% CI 2-sided [.094 to 3.582], Standard Error of Mean .539

19. Secondary Outcome: Is Your Child Able to Take Part in Hobbies or Leisure Activities?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 34 | 25
score on a scale | 2.82 (.94) | 3.28 (.89)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .673, Chi-squared; Odds Ratio (OR) = .688, 95% CI 2-sided [.121 to 3.90], Standard Error of Mean .609

20. Secondary Outcome: Is Your Child Able to Feel Independent?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 40 | 22
score on a scale | 3.13 (1.09) | 3.27 (1.03)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .544, Chi-squared; Odds Ratio (OR) = .674, 95% CI 2-sided [.189 to 2.406], Standard Error of Mean .438

21. Secondary Outcome: Has the Vest or Dressing Been Easy to Use?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 39 | 30
score on a scale | 3.54 (.72) | 3.2 (.89)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .464, Chi-squared; Odds Ratio (OR) = 1.88, 95% CI 2-sided [.345 to 10.278], Standard Error of Mean 1.631

22. Secondary Outcome: Has the Vest or Dressing Been Comfortable to Wear?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 38 | 26
score on a scale | 3 (1.07) | 2.15 (1.16)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .090, Chi-squared; Odds Ratio (OR) = 5.595, 95% CI 2-sided [.766 to 40.854], Standard Error of Mean 5.675

23. Secondary Outcome: Has the Vest or Dressing Kept You Child's Central Line Safe?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 38 | 29
score on a scale | 3.26 (.98) | 3.45 (.74)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .991, Chi-squared; Odds Ratio (OR) = .987, 95% CI 2-sided [.107 to 9.114], Standard Error of Mean 1.119

24. Secondary Outcome: Has the Vest or Dressing Prevented Your Child From Tampering With or Touching the Central Line?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 38 | 30
score on a scale | 3.16 (1.15) | 2.7 (1.15)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .223, Chi-squared; Odds Ratio (OR) = 4.239, 95% CI 2-sided [.415 to 43.326], Standard Error of Mean 5.027

25. Secondary Outcome: Has the Vest or Dressing Enabled Your Child to be More Active?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 38 | 27
score on a scale | 2.84 (1.17) | 2.67 (1.24)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .488, Chi-squared; Odds Ratio (OR) = 2.199, 95% CI 2-sided [.238 to 20.348], Standard Error of Mean 2.496

26. Secondary Outcome: Has the Presence of a Central Line Affected Their Body Image?
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 39 | 24
score on a scale | 1.72 (1.09) | 2.71 (1.33)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .018, Chi-squared; Odds Ratio (OR) = .177, 95% CI 2-sided [.0424 to .743], Standard Error of Mean .129

27. Secondary Outcome: How Would You Rate Your Child's Quality of Life on a Scale of 1 to 10?
Description: Survey modified from Baxter Scale of Quality of Life. These surveys were completed by family members or patients. Responses were recorded as a likert scale from 1-10 with 1 being very bad, 10 being very good. Quality of life data was recorded using ordinal scales. Therefore, we compared responses to individual questions between the dressing group and vest group using ordinal logistic regression, adjusting for clustering of responses within a participant. We present the mean and standard deviation for all responses as well as the ordinal odds ratio and 95% confidence intervals for a unit change in response level for each question.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 40 | 32
score on a scale | 9.16 (1.04) | 8.28 (1.78)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .269, Chi-squared; Odds Ratio (OR) = 3.688, 95% CI 2-sided [.364 to 37.379], Standard Error of Mean 4.358

28. Secondary Outcome: How Would You Rate Your Child's Ability to Cope With Day to Day Activities?
Description: Survey modified from Baxter Scale of Quality of Life. These surveys were completed by family members or patients. Responses were recorded as a likert scale from -5 to 5 with -5 being very bad, 5 being very well. Quality of life data was recorded using ordinal scales. Therefore, we compared responses to individual questions between the dressing group and vest group using ordinal logistic regression, adjusting for clustering of responses within a participant. We present the mean and standard deviation for all responses as well as the ordinal odds ratio and 95% confidence intervals for a unit change in response level for each question.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 43 | 32
score on a scale | 4.23 (1.41) | 3.5 (1.87)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .108, Chi-squared; Odds Ratio (OR) = 4.251, 95% CI 2-sided [.728 to 24.84], Standard Error of Mean 3.829

29. Secondary Outcome: How Has Your Child's Quality-of-life Been Affected by Vest or Dressing?
Description: as for outcome 28
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 41 | 32
score on a scale | 3.17 (2.34) | 1.5 (2.38)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .113, Chi-squared; Odds Ratio (OR) = 3.658, 95% CI 2-sided [.737 to 18.157], Standard Error of Mean 2.99

30. Secondary Outcome: How Has Your Child's Quality-of-life Been Affected by Their Underlying Illness?
Description: as for outcome 28
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Total Responses
Arm/Group | Device | Traditional Securement Dressing
Number analyzed (Participants) | 11 | 10
Number analyzed (Total Responses) | 44 | 32
score on a scale | 2.2 (2.86) | .59 (2.72)
Statistical Analysis 1: Comparison: Device vs Traditional Securement Dressing; Test type: Superiority; p = .049, Chi-squared; Odds Ratio (OR) = 2.495, 95% CI 2-sided [1.004 to 6.202], Standard Error of Mean 1.156

ADVERSE EVENTS:
Time Frame: 1 year from enrollment
Arm/Group | Device | Traditional Securement Dressing
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

LIMITATIONS AND CAVEATS:
Limitations include small sample size, loss of follow up and poor compliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT04522778/Prot_SAP_000.pdf